CLINICAL TRIAL: NCT01908361
Title: Hybrid Approach to Unilateral vs. Bilateral Upper Limb Rehabilitation in Subacute and Chronic Stroke
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 02-M04-022
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Cerebrovascular Accident
Keywords: comparative efficacy research; combination therapy; neurorehabilitation; robotic rehabilitation; restraint therapy
MeSH Terms: conditions — Stroke | interventions — serum P-component; Methods; glycine N-choloyltransferase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Unilateral Hybrid (InMotion3 plus CIT) Intervention (Experimental): Participants will receive 3 weeks of robot-assisted therapy (RT) using the InMotion3 Wrist Robot, followed by 3 weeks of CIT training.
  Interventions: Behavioral: Unilateral Hybrid (InMotion3 plus CIT) Intervention
- Bilateral Hybrid (BMT plus BAT) Intervention (Experimental): Participants in this bilateral treatment group will receive 3 weeks of RT using the Bi-Manu-Track (BMT) robot (Reha-Stim Co., Berlin, Germany), followed by 3 weeks of therapist-based BAT.
  Interventions: Behavioral: Bilateral Hybrid (BMT plus BAT) Intervention
- Conventional Rehabilitation (CR) (Active Comparator): The CR intervention will be designed to match the duration and intensity of the hybrid interventions.
  Interventions: Behavioral: Conventional Rehabilitation

INTERVENTIONS:
Behavioral: Unilateral Hybrid (InMotion3 plus CIT) Intervention — During the 3-week InMotion3 period, participants will receive 5 minutes of muscle tone normalization preparation and passive range of motion, then 85 minutes of training using the InMotion3 robot. The participants will practice about 5 to 8 minutes of passive, 30 to 35 minutes of assisted-active, and 5 to 8 minutes of active motions in wrist and forearm, respectively.
  During the 3-week CIT period, participants will receive intensive training of the affected UL in functional tasks with behavioral shaping for 1.5 hours/weekday and will be asked to wear a mitt to restrict the unaffected UL for 6 hours daily. The shaping techniques will involve individualized task selection, graded task difficulty, verbal feedback, prompting, physical assistance with movements, and modeling. Caregivers will use daily logs to document hours of mitt wearing outside the one-on-one intervention sessions.
  Arms: Unilateral Hybrid (InMotion3 plus CIT) Intervention
Behavioral: Bilateral Hybrid (BMT plus BAT) Intervention — During the 3-week BMT period, patients will play a simple computer game (e.g., picking up apples) that tracks patient movements to provide instant visual feedback. The therapist will also provide verbal feedback. In each training session, the patient will practice 600 to 800 repetitions of passive-passive mode for 15 minutes, 600 to 800 repetitions of active-passive mode for 15 to 20 minutes, and 150 to 200 repetitions of active-active mode for 5 minutes, respectively, for the forearm pronation-supination and the wrist flexion-extension.
  During the 3-week BAT period, participants will receive training in tasks focusing on bilateral symmetric or alternating movements of both ULs, such as lifting two cups, picking up two pegs, grasping and releasing two towels, and wiping the table with both hands.
  Arms: Bilateral Hybrid (BMT plus BAT) Intervention
Behavioral: Conventional Rehabilitation — Participants in CR group will receive therapist-mediated functional tasks training based on neurodevelopmental techniques with emphasis on functional tasks and muscle strengthening that will involve (1) active/passive range of motions, abnormal muscle tone/reflex inhibition techniques (such as stretching and/or weight bearing), and strengthening of affected arm for 15 to 20 minutes, (2) functional tasks for training fine motor or manual dexterity for 20 minutes, and (3) activities of daily living or functional tasks involving gross motor activities, coordination tasks, transition, mobility, and posture/balance for 15 to 20 minutes. The activities will be individualized according to the level of impairment and the needs of the patients.
  Other Names: CR
  Arms: Conventional Rehabilitation (CR)

SUMMARY:
In the unilateral vs. bilateral hybrid rehabilitation trials, we will conduct two separate clinical trials: one to recruit subacute stroke patients and another to recruit chronic stroke patients. The two trials will have identical study designs and interventions. The overall goal of this research project is to provide scientific evidence of the treatment effects of unilateral and bilateral hybrid therapies in subacute and chronic stroke patients and thus to contribute to evidence-based stroke rehabilitation and translational research for neurorehabilitation.

DETAILED DESCRIPTION:
The first aim of the project will be to compare treatment effects between hybrid rehabilitation and conventional rehabilitations (CR) on motor function, daily functions, mobility, quality of life, and kinematic variables. We hypothesize that patients receiving hybrid rehabilitation will gain more recovery than patients receiving CR in proximal (e.g., motor function) and in distal outcomes (e.g., quality of life) and that patients in the hybrid rehabilitation groups will show more genuine upper extremity motor recovery than those in conventional rehabilitation groups, as indicated by kinematic measures.

The second aim will be to examine the comparative treatment effects between unilateral hybrid and bilateral hybrid rehabilitation on various aspects of outcomes. We hypothesize that the unilateral group will improve more on outcomes associated with distal upper limb (UL) control and that the bilateral rehabilitation group will improve more on outcomes associated with proximal UL control.

Third, we will collect biomarker indexes before and after the interventions to monitor the changes of oxidative stress and inflammatory levels.

ELIGIBILITY:
Inclusion Criteria:

* 1 to 6 months onset from a first-ever unilateral stroke for the subacute randomized controlled trial (RCT), and more then 6 months after onset for the chronic RCT
* minimal motor criteria to receive CIT (i.e., ≥10º wrist extension and ≥ 10º extension at the thumb and any two other digits)
* an initial FMA-UE score of 18 to 56, indicating mild to moderate and moderate to severe upper extremity motor impairment
* no excessive spasticity in any of the joints of the affected arm (shoulder, elbow, wrist, and fingers)
* able to follow instructions and perform the study tasks (Mini Mental State Examination ≥ 24)
* without upper extremity fracture within 3 months
* no participation in any rehabilitation experiments or drug studies during the study period
* willing to provide written informed consent

Exclusion Criteria:

* acute inflammatory disease
* major health problems or poor physical condition that might limit participation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Fugl-Meyer Assessment (FMA) | Baseline, 3 weeks, 6 weeks, and 18 weeks
  The upper-extremity subscale of the FMA will be used to assess motor impairment. The 33 upper limb items measure the movement and reflexes of the shoulder/elbow/forearm, wrist, hand, and coordination/speed. They are scored on a 3-point ordinal scale (0-cannot perform, 1-performs partially, 2-performs fully). The maximum score is 66, indicating optimal recovery. The sub-score of a proximal shoulder/elbow (FMA s/e: 0-42) and a distal hand/wrist (FMA h/w: 0-24) will be also calculated to investigate the treatment effects on separate upper extremity elements. The reliability, validity, and responsiveness of the FMA in stroke patients have been shown to be good.
Change in Wolf Motor Function Test (WMFT) | Baseline, 3 weeks, 6 weeks, and 18 weeks
  The WMFT was originally designed to assess the effects of CIT on the return of arm function for stroke and traumatic brain injury. The assessment requires the participant to perform 15 function-based and 2 strength-based tasks. The tasks are averaged to produce a score in seconds that ranges from 0 to 120 seconds. For functional ability scoring, we used a 6-point ordinal scale where 0 indicates "does not attempt with the involved arm" and 5 indicates "arm does participate; movement appears to be normal." The clinimetrics of the WMFT has been ascertained in stroke patients.

SECONDARY OUTCOMES:
Change in MyotonPro | Baseline, 3 weeks, 6 weeks, and 18 weeks
  The MyotonPRO represents a noninvasive way to characterize the viscoelastic properties of skeletal muscle in vivo. Three measurement parameters in the MyotonPRO: F - Frequency, Hz, characterizes muscle tone; D - Decrement, characterizes muscle elasticity; S - Stiffness, N/m, characterizes muscle stiffness. The working principles of the MyotonPRO are as follows: the testing end of the MyotonPRO will be placed perpendicular to the skin surface above the muscle to be measured, a brief mechanical impulse will be applied, shortly followed by a quick release to the muscle through an acceleration probe, and the damped oscillations of the muscle response will be recorded by the acceleration transducer at the testing end of the device. The oscillation graph creates during the measurement expresses the acceleration of the testing end.
Change in 10-Meter Walk Test (10MWT) | Baseline, 3 weeks, 6 weeks, and 18 weeks
  The 10MWT assess mobility function by measuring the time and the numbers of strides required to walk 10 meters under two conditions: (1) with the self-pace of each participant (self-pace); (2) with the speed that the participants walked as soon as possible. The velocity and stride length of the participant are calculated. Research has validated the 10MWT in measuring mobility in stroke.
Change in Actigraphy | Baseline, 3 weeks, 6 weeks, and 18 weeks
  The activity monitors will be used to provide a direct and objective measure of the amount of the impaired arm movement outside the laboratory. This measure, quantitatively recording the amount of activity in free-living conditions, will be used to reflect increase in the amount of affected arm use over time. The participants will be asked to wear an activity monitor, Actigraphy (Ambulatory Monitoring Inc., New York), on each wrist for 3 consecutive days to measure what amount they actually do in their daily life before and immediately after treatment. The Actigraphy can be attached to the subject's limb and measures the motion of that limb through an accelerometer. In this project, acceleration will be sampled at 10 Hz and summed over a user-specified epoch. The recording epoch will be 2 seconds; recording capacity will be approximately 72 hours. The ratio of affected to non-affected arm movement is a reliable and valid real-life measure of treatment outcome.
Change in Functional Independence Measure (FIM) | Baseline, 3 weeks, 6 weeks, and 18 weeks
  The FIM consists of 18 items grouped into 6 subscales measuring self-care, sphincter control, transfer, locomotion, communication, and social cognition ability. Each item is rated from 1 to 7 (maximum score 126) based on the required level of assistance to perform the tasks (e.g., 1-complete assistance and 7-complete independence). A higher score on any subscale indicates a less disability. The FIM has been shown to have good inter-rater reliability, construct validity, and discriminant validity.
Change in Motor Activity Log (MAL) | Baseline, 3 weeks, 6 weeks, and 18 weeks
  The MAL consists of 30 structured questions to interview how the patients rate the frequency (amount of use subscale) and quality (quality of movement subscale) of movements while using their affected arm to accomplish each of the 30 daily activities. The score of each item ranges from 0 to 5, and the higher scores indicate more frequently used or higher quality of movements. The summary score is the mean of the item scores. The clinimetric properties of the MAL in stroke patients have been validated.
Change in ABILHAND Questionnaire | Baseline, 3 weeks, 6 weeks, and 18 weeks
  The ABILHAND Questionnaire will be used to evaluate the ability of the UL in functional activities. It consists of 23 bimanual activities that measure subjectively perceived difficulty in performing some common activities in daily living, such as buttoning, cutting nails, and opening a bottle. The scale ranges from 0 to 3 (0 = cannot perform, 1 = performs partially or with great difficulty, 2 = performs with some difficulty, 3 = performs fully). Its reliability and construct validity has been confirmed.
Change in Nottingham Extended Activities of Daily Living Scale (NEADL) | Baseline, 3 weeks, 6 weeks, and 18 weeks
  he NEADL consists of 22 items scored on the basis of the requirement for help in performing the activity. There are four subscales (mobility, domestic, leisure and kitchen) and a total score. The scores range from 0 to 22, with higher scores representing better function. The psychometric properties of the NEADL have been validated in stroke patients.
Change in Stroke Impact Scale Version 3.0 (SIS 3.0) | Baseline, 3 weeks, 6 weeks, and 18 weeks
  The SIS 3.0 is a stroke-specific instrument of health-related quality of life. It contains 59 items measuring 8 domains (i.e., strength, hand function, activities of daily living/instrumental activities of daily living, mobility, communication, emotion. memory and thinking and participation) with a single item assessing perceived overall recovery from stroke. Items are rated on a 5-point Likert scale with lower scores indicating greater difficulty in task completion during the past week. The reliability, validity, and responsiveness have been shown to be satisfactory in stroke patients.
Change in Physiologic Response Measures (Biomarkers) | Baseline, 3 weeks, 6 weeks, and 18 weeks
  Proinflammatory markers and anti-inflammatory markers will be used to monitor changes in inflammation. Proinflammatory markers include C-reactive protein (CRP), tumor necrosis factor-α (TNF-α), interleukin (IL)-1α, and IL-6. Anti-inflammatory markers include IL-10 and transforming growth factor-β1 (TGF-β1). Oxidative stress and antioxidative markers will be used to monitor the changes on oxidative stress. Oxidative stress makers include 8-hydroxy-2-deoxyguanosine (8-OHdG) and F2-isoprostances. The antioxidants will include antioxidants superoxide dismutase (SOD) and glutathione peroxidase (GPx). We have no directional hypotheses regarding the changes of biomarkers because of its early stage in stroke rehabilitation research.
Change in Kinematic analysis | Baseline, 3 weeks, 6 weeks, and 18 weeks
  The kinematic analysis will involve unilateral and bilateral tasks, in which the participants will be asked to perform by using the affected upper limb or both upper limb simultaneously. A motion analysis system with 7 cameras (VICON MX 30d, Oxford Metrics Inc., Oxford, UK) will be used to capture the motion of arm (s) in kinematic testing. The markers will be attached on the styloid processes of the ulna. Depending on the unilateral or bilateral tasks, the makers will be placed on the affected arm or the both arms, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Keh-chung Lin, ScD, Principal Investigator — School of Occupational Therapy, College of Medicine, National Taiwan University, Taiwan; Yi-shiung Horng, PhD, Principal Investigator — Buddhist Tzu Chi General Hospital Taipei Branch
Locations (1):
- Buddhist Tzu Chi General Hospital Taipei Branch, New Taipei City, Taiwan, Taiwan